CLINICAL TRIAL: NCT03785652
Title: Multicenter,Randomized,Double-blind,Placebo,Parallel-controlled,Dose-Finding Clinical Trial to Evaluate the Efficacy and Safety of LY03005 Extended-release Tablets in the Treatment of Major Depressive Disorder (MDD)
Brief Title: Dose-Finding Clinical Trial to Evaluate the Efficacy and Safety of LY03005 Extended-release Tablets in the Treatment of Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Shandong Luye Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY03005-CHN-204
Record Dates: First submitted 2018-12-17; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY03005 extended-release tablets (Experimental): LY03005 extended-release tablets at 4 doses 40 mg, 80mg, 120mg or 160mg
  Interventions: Drug: LY03005 extended-release tablets 40 mg; Drug: LY03005 extended-release tablets 80 mg group; Drug: LY03005 extended-release tablets 120 mg group; Drug: LY03005 extended-release tablets 160 mg group
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: LY03005 extended-release tablets 40 mg — LY03005 extended-release tablets 40 mg group :40mg/day，orally once a day, at a regular morning time on an empty stomach or after breakfas
  Arms: LY03005 extended-release tablets
Drug: LY03005 extended-release tablets 80 mg group — LY03005 extended-release tablets 80 mg group :
  80mg/day，orally once a day, at a regular morning time on an empty stomach or after breakfast
  Arms: LY03005 extended-release tablets
Drug: LY03005 extended-release tablets 120 mg group — LY03005 extended-release tablets 120 mg group :
  120mg/day，orally once a day, at a regular morning time on an empty stomach or after breakfast
  Arms: LY03005 extended-release tablets
Drug: LY03005 extended-release tablets 160 mg group — LY03005 extended-release tablets 160 mg group :
  160mg/day，orally once a day, at a regular morning time on an empty stomach or after breakfast
  Arms: LY03005 extended-release tablets
Drug: Placebo group — Placebo group :
  Placebo ，orally once a day, at a regular morning time on an empty stomach or after breakfast
  Arms: Placebo

SUMMARY:
This study was a multicenter, randomized, double-blind, placebo, parallel-controlled, dose-finding Phase II clinical trial to find the optimal dose of LY03005 Extended-release Tablets for the treatment of MDD and to evaluate the preliminary efficacy and safety, providing a basis for the design of phase III clinical trials and the determination of dosing regimens.

DETAILED DESCRIPTION:
The study consisted of two periods: a screening and washout period of 2 weeks (recommended 8 days) and a double-blind treatment period (6 weeks). The first period is the screening and washing period, the longest is 14 days and the shortest is 8 days (recommended 8 days), in which the enrolled MDD subjects will start a one-week placebo wash period and receive prescribed a placebo, 2 pills once a day for 7 consecutive days. The second period was a double-blind treatment period of 6 weeks. After the placebo washout period, 260 enrolled subjects were randomized into one of 5 study groups in the 1:1:1:1:1 ratio, 4 LY03005 Extended-release Tablets treatment groups with different dose or 1 placebo group. Subjects were given investigatory drug or placebo according to the protocol, 4 pills once a day and followed up at the end of 1, 2, 4 and 6 weeks.

Effectiveness of the investigational drug was evaluated using 17 Hamilton Depression Scale (HAM-D17), Montgomery-Asberg Depression Scale (MADRS), Hamilton Anxiety Scale (HAMA), Clinical Global Impression Scale (CGI) and Visual Analog Scale-Pain intensity (VAS-PI) scores. Safety of the treatment was evaluated by adverse events, vital signs, laboratory measurements (blood routine, urine routine, blood biochemistry and serology), 12-lead ECG, physical examination, the Arizona Sexual Experience Scale (ASEX) and the Columbia-Suicide Severity Rating Scale (C-SSRS) scores.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 to 65 years subjects from outpatient or inpatient;
2. Subjects who meet the diagnostic criteria for MDD in DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders, 4th Edition) with either single or recurrent episodes (296.2/296.3) without psychotic characteristics;
3. Total scores of 17-item Hamilton Depression Scale (HAM-D17) ≥ 20 points at screening and baseline visits；
4. First item (depressive mood) score of HAM-D17 scale ≥ 2 points at screening and baseline visits;
5. Clinical global impression scale-disease severity (CGI-S) score ≥ 4 points at screening and baseline visits;
6. At screening and baseline, women of childbearing age (e.g., women who have not undergone surgical sterilization or less than one year after menopause) have a urine negative pregnancy test result. Male and female subjects of childbearing age agree to take effective contraceptive measures during the entire study period and at least 28 days after the last dose of investigatory drug;
7. Subjects voluntarily participate in the trial by signing the informed consent form and are able to follow the schedule in the protocol for visits, treatment, laboratory tests and other research procedures.

Exclusion Criteria:

1. Allergic or known to be allergic to venlafaxine and desvenlafaxine;
2. MDD subjects who were not responsive to the previous venlafaxine treatment with sufficient amount and duration or TRD, to at least two different mechanisms of action antidepressants with adequate amount and duration in the past;
3. Total scores of HAM-D17 scale at baseline was decreased ≥25% compared with the one at screening;
4. There is a clear suicide attempt or behavior and score of the 3rd item (suicidal thought) in HAM-D17 total scale ≥ 3 points;
5. Gestational and lactating women or the subjects of childbearing age who do not take effective contraception or who do not agree to continue using contraception within 28 days of the last dose;
6. Suppressed subjects who also meet other diagnoses on the DSM-IV-TR axis I or received the treatment for such diagnoses (including current or previous diagnosis of anorexia nervosa or bulimia nervosa), or was diagnosed as dysthymia in the past 2 years;
7. MDD secondary to other mental illnesses or physical illnesses;
8. Those with a history of seizures (except for convulsions caused by febrile seizures in children);
9. Those receiving electroconvulsive therapy (ECT) within 3 months prior to screening or according to the investigator's judgment that ECT is currently required; Those who have received systematic psychotherapy (interpersonal relationship therapy, dynamic therapy, cognitive behavioral therapy) within 3 months prior to screening；Those who have received transcranial magnetic stimulation (TMS) within 3 months prior to screening, or have received light therapy within 2 weeks prior to screening;
10. Subjects who have regularly taken anti-depressants within 2 weeks prior to screening, and have stopped the anti-depressants less than 2 weeks or psychotropic drugs for less than 7 half-lives prior to study randomization (monoamine oxidase inhibitor for at least 2 weeks, fluoxetine for at least 1 month);
11. Subjects who have seriously unstable cardiovascular, liver, kidneys, blood, endocrine and other physical diseases or a medical history;
12. Hypertensive patients with poor blood pressure control (SBP≥140 mmHg or DBP≥90 mmHg at screening and baseline);
13. There is a history of gastrointestinal disease known to interfere with drug absorption or excretion or a history of surgery known to interfere with drug absorption or excretion;
14. A history of increased intra-ocular pressure or narrow-angle glaucoma;
15. Clinically significant abnormalities based in investigators judgment during screening (for example, such as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is 1.5 times higher than upper limit of normal range; creatinine (Cr) is higher than the upper limit of normal ranges and clinical significant abnormal thyroid function);
16. Electrocardiogram (ECG) abnormalities are clinically significant at screening and the investigators believe that it is inappropriate for the subjects to be enrolled, such as QTc interval ≥450 ms for male and QTc interval ≥460 ms for female;
17. Those who have participated in other clinical trials within 3 months prior to screening;
18. Those with serious acute or chronic diseases, mental illnesses or clinically significant abnormalities in laboratory tests, of which investigators believe that the subjects are not suitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale | 8 weeks
  Changes from baseline in the total score of 17 items of Hamilton Depression Scale (HAM-D17) at the end of treatment

SECONDARY OUTCOMES:
Montgomery- Åsberg Depression Rating Scale(MADRS) | 8 Weeks
  Changes from baseline in the 10-items Montgomery- Åsberg Depression Rating Scale(MADRS) total scores at the end of treatment;
Clinical Global Impression Scale - improvement (CGI-I) | 8 Weeks
  Changes in the Clinical Global Impression Scale - improvement (CGI-I) scores at the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Approval Letter of Ethics Committee of The Sixth Hospital of Peking University, Haidian District,, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No